CLINICAL TRIAL: NCT06655857
Title: Interventions for Promoting Kidney Transplant Empowerment
Acronym: INSPIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lili Chan, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GCO 22-1921; U01DK137259 (NIH)
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Kidney Transplant Waitlisting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Community Health Worker and Intervention Providers-Assisted Kidney Transplant Support (Other): Participants will receive assignment to a community health worker who will educate them on the kidney transplant process, assist them through the kidney transplant process and connect them with any necessary social services.
  Interventions: Other: Community Health Worker Assistance; Other: Intervention Providers
- Usual Care (Other): Participants will receive usual care and at the end of the study will receive education, and work with CHWs in a more limited capacity. Control clinicians will receive the education intervention.
  Interventions: Other: Usual Care; Other: Community Health Worker Assistance; Other: Intervention Providers

INTERVENTIONS:
Other: Usual Care — Participants are provided care as usual. Clinicians (CKD, HD, KTx) will educate participants on the kidney transplant process. Clinician will receive the education intervention to provide participants at study end.
  Arms: Usual Care
Other: Community Health Worker Assistance — Community health worker will address unmet social needs and participant symptoms through evaluations and intake to clinical and community services
Other: Intervention Providers — Intervention providers will receive education, which will include training on working with CHWs, reducing bias in clinical decision-making, and increasing affirming/reducing stigmatizing language in electronic health records (EHRs).

SUMMARY:
This is a cluster randomized controlled clinical trial evaluating the effect of community health workers (CHWs) and provider education on kidney transplant (KTx) waitlisting compared to usual care (waitlist control). CKD/HD providers will be randomized to intervention or control, and all patients with the same providers will be in the same randomization group. CHWs will address unmet social needs and patient symptoms through evaluations and linkage to clinical and community services. Intervention providers will receive education, which will include training on working with CHWs, reducing bias in clinical decision-making, and increasing affirming/reducing stigmatizing language in electronic health records (EHRs).

ELIGIBILITY:
Inclusion Criteria:

* Patient inclusion:

  * Provision of signed and dated informed consent from the patient.
  * Stated willingness to comply with all study procedures and availability for the duration of the study.
  * Age 18 - 75 years
  * eGFR≤20 mL/min/1.73m2 or on maintenance in-center HD.
  * Receive kidney care at Mount Sinai, Einstein, Bellevue Hospital, NYU, or hemodialysis at a participating HD Center.
  * Community dwelling (i.e., not in a nursing home, currently incarcerated).
  * Speak English and/or Spanish.
* Provider Inclusion:

  * Provision of signed and dated informed consent from the nephrologist.
  * Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Patient Exclusion:

  * Absolute contraindications to KTx:

    * Self-reported or documented diagnosis of dementia, or inability to understand the study and complete informed consent. When the participant's understanding is unclear, the CRC will use a modified MOCA screener to determine eligibility.
    * Active malignancy (excluding local non-melanoma skin cancer, renal cell carcinoma <5 cm, early thyroid cancer, and prostate cancer GS≤6).
    * Pregnancy (can be re-evaluated post-delivery).
    * Active infection. Patients excluded due to active infection will be evaluated at 30 days or after completing full treatment (whichever is later) to determine eligibility. Examples of active infection include:

      * Positive cultures or radiographic evidence of infection
      * Infected intravascular devices, such as tunneled catheters and pacemakers
      * Active histoplasmosis, cryptococcosis, tuberculosis (TB), and nontuberculous mycobacteria
  * Previously evaluated by KTx and not listed for specific medical reasons.
  * Patients previously evaluated and not listed will be carefully reviewed by site PI for eligibility
  * Already listed for KTx.
  * Patients on other types of dialysis other than in-center hemodialysis.
  * Self-identify as already engaged with a CHW at participating sites to address unmet social needs.
  * Planning to move out of the greater NY area in the next 1 year.
* Provider Exclusion:

  * Planning to leave their respective institutions in the next 1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to completion of kidney transplant waitlisting evaluation | Baseline, and then every 6 months up to 2 years
  Patient medical records will be reviewed, and the patient will be asked directly for the status of their kidney transplant evaluation.

SECONDARY OUTCOMES:
Accountable Health Communities Health-Related Social Needs Screening Tool (AHC-HRSN) | Baseline, and then every 6 months up to 2 years
  The AHC-HRSN is a 10-item screening tool designed to help providers identify patients' needs across five core domains: Housing Instability, Food Insecurity, Transportation Problems, Interpersonal Safety, and Utility Help needs. Each item is scored using a Yes/No response format. If a patient answers "Yes" to any of the items, they are considered to have screened positive for a safety need.
Discrimination in Medical Settings (DMS) | Baseline, and 12 months after first study visit
  The Discrimination in Medical Settings (DMS) Scale is a modified version of the EDS that has been previously used to study perceived discrimination in medical settings, among patients with a range of clinical conditions. Responses to each of the 7 items are assessed with a 5-point Likert scale. Scores range from 7-35. Higher scores indicate higher frequencies of experiences with everyday mistreatment.
Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v1.2 | Baseline, and 12 months after first study visit
  The Patient Reported Outcomes Measurement Information System (PROMIS) Scale v1.2 - Global Health is a patient reported measure of physical, mental and social health. Items query general health, quality of life, physical health, mental health, satisfaction with discretionary social activities, carrying out every day physical activities, pain, fatigue, satisfaction with social roles, and emotional problems. For scoring, Item-levels are scored numerically for an individual's response to each question. Responses to each of the items are assessed with a 5-point Likert scale. Raw scores range from 7-35. Higher scores indicate higher presence of symptom.
Initiation of KTx process | Baseline, and 12 months after first study visit
  Will measure whether or not the patient started the kidney transplant process. Patient medical records will be reviewed to see if there is a date available and/or ask the patient directly. A response of yes/no will be recorded.
Binary outcome of patient being KTx waitlisted or not by year 1 post enrollment | Baseline, and 12 months after first study visit
  Will measure whether or not the patient has been waitlisted for a kidney transplant at 1 year out from being enrolled in the trial. Patient medical records will be reviewed to see if there is a date available and/or ask the patient directly for confirmation. A response of yes/no will be recorded.
Binary outcome of patient being KTx waitlisted or not by year 2 post enrollment | Baseline, and then every 6 months up to 2 years after patients first study visit
  Will measure whether or not the patient has been waitlisted for a kidney transplant at 2 years out from being enrolled in the trial. Patient medical records will be reviewed to see if there is a date available and/or ask the patient directly for confirmation. A response of yes/no will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lili Chan, Principal Investigator — Ichan School of Medicine at Mount Sinai Hospital
Locations (3):
- United States (3):
  - NYU Langone Health, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Montefiore Einstein, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No
All data will be deidentified for analysis